CLINICAL TRIAL: NCT00362284
Title: Expanded Counseling and Support for Adult Children Caring for Parents With Alzheimer's Disease or Similar Disorders
Brief Title: Comprehensive Support for Alzheimer's Disease Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: H13355B; R01AG022066 (NIH)
Record Dates: First submitted 2006-08-08; First posted 2006-08-09 (Estimated); Last update posted 2022-02-11 (Actual); Status verified 2022-02

CONDITIONS: Caregivers; Stress; Depression
Keywords: Alzheimer's disease; coping; quality of life; caregiving
MeSH Terms: conditions — Depression; Alzheimer Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NYUCI-AC group (Experimental): Adult children in this arm received the NYUCI-AC intervention, which consisted of 6 individual and family counseling sessions, the offering of an adult child specific support group, and the provision of ad hoc, or ongoing, consultation throughout the duration of participation.
  Interventions: Behavioral: NYUCI-AC
- Usual care control (No Intervention): Adult children randomly assigned to the usual care control did not receive the NYUCI-AC intervention. If they were in crisis or required support, the NYUCI-AC counselors provided information and referral on an as-needed basis.

INTERVENTIONS:
Behavioral: NYUCI-AC — Approximately six individual and family consultation sessions (2 individual, 3 family, 1 individual) within the first 4 months with adult child caregivers and/or their family members; support group participation (recommended at least once a month) after the completion of the individual and family consultation sessions for the duration of the project (up to 3 years after the intake interview); ad hoc consultation (ongoing in-person, telephone, or email support on an as-needed basis) for the duration of the project (up to 3 years after the intake interview); New York University Caregiver Intervention
  Arms: NYUCI-AC group

SUMMARY:
The purpose of this study is to determine the effectiveness of a comprehensive counseling and support intervention for people who care for parents with Alzheimer's disease (AD) or other dementias on outcomes such as stress, depression and ability to postpone or avoid nursing home placement.

DETAILED DESCRIPTION:
Although a range of studies have examined the stress and depression of family caregivers of persons suffering from dementia, the effectiveness of psychosocial interventions to assist caregiving families and their disabled elderly relatives is uncertain. The comprehensive support protocol to be implemented, the Enhanced Counseling and Support (ECS) program, has been successfully implemented at the Silberstein Aging and Dementia Research Center of New York University School of Medicine (NYU-ADRC) over the past 19 years. However, the initial evaluation of the ECS was limited to a single geographic area (New York City proper) and a specific type of dementia caregiver (spouses).

The specific aims of this 4-year project are as follows: 1) Examine whether the ECS can achieve positive outcomes for adult child caregivers. Few psychosocial interventions are directed specifically at adult child caregivers, and evaluating the ECS in adult child caregiving situations, which few studies have done, will further demonstrate the effectiveness of this program and add considerably to the AD caregiver intervention literature; and 2) Determine if the ECS, an intervention of proven efficacy for AD caregivers in a northern U.S. urban community (New York City), will also be effective in alleviating negative outcomes among AD caregivers at a Midwestern project site. The study will ascertain whether the comprehensive support program developed at NYU is generalizable to caregivers from areas other than the New York City area and leads to similar benefits that are maintained over long periods of time (i.e., up to 3.5 years).

In order to accomplish the specific aims of the project, the following study hypotheses have been proposed:

1. Adult child caregivers in the treatment conditions of the University of Minnesota (UM) and NYU-ADRC will report similar decreases on measures of stress when compared to usual-contact controls;
2. Adult child caregivers in the intervention conditions at both sites will develop improved social support resources and experience significantly greater decreases of family conflict in a similar manner;
3. Adult child caregivers in the treatment conditions at UM and NYU-ADRC will report similar decreases on global measures of psychological distress, such as depression. Similarly, treatment caregivers will report greater increases in subjective health than their counterparts in the usual-contact control; and
4. Membership in the treatment condition of the ECS and its benefits (e.g., increased social support, decreased stress) will lead to delayed institutionalization (e.g., nursing home placement) of care recipients at the UM and NYU-ADC sites.

ELIGIBILITY:
Inclusion Criteria:

* Participant (i.e., adult child) must be the 'primary' caregiver of the patient with a diagnosis of dementia (i.e., the first person called if the patient is in need of help) at the time of the baseline interview
* Must be a daughter, son, daughter-in-law, or son-in-law of the patient
* Patient must live in the community (i.e., at home, with the caregiver, with other relatives)
* Sees the individual with dementia once a week or more

Exclusion Criteria:

* Unable to understand or speak English comfortably
* Inadequate hearing
* Unwilling to participate in the study or sign the consent form
* Suffered from or received treatment for an emotional or psychological disorder, such as depression, anxiety, or some other type of psychotic episode, within the past 6 months
* Not physically able to participate
* Received counseling for problems arising as a caregiver

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2005-09; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Care recipient nursing home/institutional placement | baseline, 4, 8, 12, and 18 months; 24, 30, 36 months if possible
  Adult child caregivers self-reported whether the care recipient was admitted to a residential care setting and the date of admission.
Caregiver emotional stress | baseline, 4, 8, 12, and 18 months; 24, 30, 36 months if possible
  Measures of role captivity, role overload, and general perceived stress.
caregiver depression | baseline, 4, 8, 12, and 18 months; 24, 30, 36 months if possible
  The Geriatric Depression Scale.
caregiver social support | baseline, 4, 8, 12, and 18 months; 24, 30, 36 months if possible
  Three single items that measured perceptions of support received by the adult child caregiver.

SECONDARY OUTCOMES:
Caregiver subjective health | baseline, 4, 8, 12, and 18 months; 24, 30, 36 months if possible
  Single item self-reported health as well as measures derived from the OARS.
secondary stressors | baseline, 4, 8, 12, and 18 months; 24, 30, 36 months if possible
  Measures of family and role conflict.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph E. Gaugler, PhD, Principal Investigator — University of Minnesota, Center on Aging, Center for Gerontological Nursing, School of Nursing; Mary Mittelman, DrPH, Principal Investigator — Silberstein Institute for Aging and Dementia, Department of Psychiatry, NYU School of Medicine
Locations (2):
- United States (2):
  - University of Minnesota, School of Nursing, 6-150 Weaver-Densford Hall, Minneapolis, Minnesota
  - Silberstein Institute for Aging and Dementia, Department of Psychiatry, NYU School of Medicine, New York, New York

REFERENCES:
- [Background] Gaugler JE, Reese M, Mittelman MS. Process Evaluation of the NYU Caregiver Intervention-Adult Child. Gerontologist. 2018 Mar 19;58(2):e107-e117. doi: 10.1093/geront/gnx048. PMID 29562359
- [Result] Gaugler JE, Reese M, Mittelman MS. Effects of the NYU caregiver intervention-adult child on residential care placement. Gerontologist. 2013 Dec;53(6):985-97. doi: 10.1093/geront/gns193. Epub 2013 Jan 20. PMID 23339050
- [Result] Gaugler JE, Reese M, Mittelman MS. Effects of the Minnesota Adaptation of the NYU Caregiver Intervention on Primary Subjective Stress of Adult Child Caregivers of Persons With Dementia. Gerontologist. 2016 Jun;56(3):461-74. doi: 10.1093/geront/gnu125. Epub 2015 Jan 27. PMID 25628299
- [Result] Gaugler JE, Reese M, Mittelman MS. Effects of the Minnesota Adaptation of the NYU Caregiver Intervention on Depressive Symptoms and Quality of Life for Adult Child Caregivers of Persons with Dementia. Am J Geriatr Psychiatry. 2015 Nov;23(11):1179-92. doi: 10.1016/j.jagp.2015.06.007. Epub 2015 Jun 25. PMID 26238226
- [Result] Gaugler JE, Reese M, Mittelman MS. The Effects of a Comprehensive Psychosocial Intervention on Secondary Stressors and Social Support for Adult Child Caregivers of Persons With Dementia. Innov Aging. 2018 Jun;2(2):igy015. doi: 10.1093/geroni/igy015. Epub 2018 Jun 22. PMID 30009268
- [Result] Albers, Elizabeth, A. (2020). A Longitudinal Analysis of the Effects of the NYU Caregiver Intervention-Adult Child on Subjective Health. Retrieved from the University of Minnesota Digital Conservancy, http://hdl.handle.net/11299/217050.